CLINICAL TRIAL: NCT01607437
Title: 10-year Follow-up After ACL Reconstruction With Howells Guide, Transtibial Drilling and Hamstrings Graft
Brief Title: Clinical Follow-up After ACL Reconstruction
Acronym: Howell
Status: Completed | Type: Observational
Sponsor: Bergen Knee Group (Other)
Responsible Party: Principal Investigator, Eivind Inderhaug, Medical Doctor, Bergen Knee Group
Other Study IDs: HowellFollowUp
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Deficiency of Anterior Cruciate Ligament; Injury of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
No former studies have done long-term evaluation on patients reconstructed with hamstrings graft, the use of Howells tibial guide and transtibial drilling of the femoral graft tunnel. The investigators aim to evaluate clinical, radiographic and subjective outcome at a minimum of 10 years after surgery. According to former published studies on alike methods, the use of transtibial drilling of the femoral graft tunnel causes an increased rotational instability of the knee. The investigators aim to map the clinical stability of this group as well as evaluating the general outcome at the long-time horizon.

DETAILED DESCRIPTION:
Patients will be invited to a clinical follow-up with x-ray of the knee, scoring of Lysholm and IKDC subjective scores, clinical examination including instrumented testing with a KT-1000. After informed consent data will be collected from patient records and stored in a secured internal database. Analysis will be done with the SPSS package.

ELIGIBILITY:
Inclusion Criteria:

- Patients reconstructed with the given technique

Exclusion Criteria:

* Patients reconstructed with other techniques
* Concomitant ligamental surgery
* Bilateral ACL injury
* Revision surgery

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients reconstructed with Howells guide, hamstrings graft and transtibial drilling at Haraldsplass Deaconess Hospital from 1999 to 2001.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Revision surgery | 10 years
  When patients have had a new ACL reconstruction of the ACL

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Inderhaug, MD, Principal Investigator — Bergen Knee Group
Locations (1):
- Haraldsplass Deaconess Hospital, Bergen, Norway